CLINICAL TRIAL: NCT03891719
Title: Correction of the Unilateral Cleft Lip Nasal Deformity Using Sliding Chondrocutaneous Flap, Caudal Septal Extension Graft and Auricular Cartilage Graft
Brief Title: Correction of the Unilateral Cleft Lip Nasal Deformity With Sliding Chondrocutaneous Flap and Autologous Cartilage Graft
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Medicine and Pharmacy at Ho Chi Minh City (Other)
Collaborators: Gia Dinh People Hospital (Other)
Responsible Party: Principal Investigator, Chuong Dinh Nguyen, MD, Principle Investigator, University of Medicine and Pharmacy at Ho Chi Minh City
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4052/QD-DHYD
Record Dates: First submitted 2019-03-24; First posted 2019-03-27 (Actual); Last update posted 2021-02-10 (Actual); Status verified 2021-02

CONDITIONS: Cleft Lip, Unilateral
Keywords: rhinoplasty; cleft lip nose; autologous cartilage graft; asian nose
MeSH Terms: conditions — Cleft Lip

STUDY DESIGN:
Intervention Model Description: we conduct a prospective analysis of 35 cases to assess difference between preoperative and postoperative nostril symmetry by using autologous cartilage graft and sliding chondrocutaneous flap
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Changes in nose symmetry (Experimental): - Direct anthropometric assessment (frontal, oblique, lateral and basal views) and three- dimensional observations of the nose preoperatively and postoperatively in order to evaluate the nostril symmetry, the angles, ratios of the nose and its relation to the face.
  Interventions: Procedure: Unilateral cleft lip rhinoplasty

INTERVENTIONS:
Procedure: Unilateral cleft lip rhinoplasty — * Perform marking with methylene blue tattoo marks
  * Inject Local anesthetic solution with epinephrine
  * Harvest auricular cartilage
  * Make the incisions parallel the lip scar, extende into the marginal incision and encompass any alar webbing. The incisions outline the entirety of the lower lateral cartilage and create sliding chondrocutaneous flap. This flap combines with reverse U incision.
  * Harvest septal bony cartilaginous unit for grafting the caudal septum and suspend the medial crural cartilages
  * Create dome symmetry at the cartilage level and reconstruct nasal tip with other grafts (shield-type tip graft, cap graft, alar batten graft)
  * Dorsal augmentation
  * Lip reconstruction and alar base repositioning.
  * Closure and repair vestibular deficiency with the reverse-U component of the chondrocutaneous flap at the alar rim.

SUMMARY:
Cleft lip and cleft palate are the most common birth defects of craniofacial development. The surgical repair of this deformity requires comprehensive management plans and well cooperating interdisciplinary cleft teams. Secondary cleft rhinoplasty remains one of the most challenging procedures and aims for restoring nostril symmetry, enhancing nasal function, and improvement of aesthetic outcomes.

DETAILED DESCRIPTION:
For the majority of cleft patients, surgeons usually delay secondary rhinoplasty to ages 14 to 16 years for females and 16 to 18 years for males until after completion of nasal growth Unilateral secondary cleft nasal deformity results from hypoplastic nasal tissue, asymmetric growth due to impaired growth, and surgical scarring. The most common deformities include caudal septal deviation, retrodisplacement and under-projection of dome, lateral slumping of the medial crus of the lower lateral cartilage, alar-columellar web, insufficiency of vestibular skin and deficiency of nasal floor. Moreover, these deformities have negative effect on human well-being and quality of life.

Despite the opinions on how to address the problems, it seems clear that repositioning and reshaping of the cleft-side cartilages is necessary for restoring form and function. In general, in order to there are two basic approaches: those techniques that move the cleft-side lower lateral cartilage from medial to lateral, and those that move the lower lateral cartilage from lateral to medial. In an effort to correct the vestibular lining deficiency, easily be adapted to combine Tajima's reverse-U incisions for treatment of alar hooding, need for other structural grafts, sliding chondrocutaneous flap offers many advantages. However, in order to improve nasal tip position or columella shape through modification of either the anterior septal and/or posterior septal angle position and to act as the fundamental attachment for sliding lower lateral cartilage, Caudal septal extension and Columellar strut graft play an important role to stabilize the nasal tip.

Besides, with the aim of making it harmonize better with other facial features, dorsal augmentation is needed for improving the shape of the nose. Selecting the optimal material continues to be a challenge. For most surgeons, an autogenous cartilage graft is the first choice in rhinoplasty because of its resistance to infection and resorption.

We assess the functional and aesthetic outcomes based on three criteria:

1. Change in nose symmetry and nasal height (Preoperative and postoperative photographic analyses)
2. Change in functional outcomes through subjective and objective measurement (Questionaire and acoustic rhinometry)
3. Change in Quality of life (Rhinoplasty Outcome Evaluation Questionaire)

ELIGIBILITY:
Inclusion Criteria:

* Patients with unilateral cleft lip deformity that was previously performed primary cheiloplasty
* No other craniofacial malformation
* Age: > 14-16 years old in female, >16-18 years old in male
* Patients with follow-up period of at least 6 months.

Exclusion Criteria:

- Patients who were suffered infection of facial structure

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2019-07-01 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2023-11 (Estimated)

PRIMARY OUTCOMES:
Assessment of nose symmetry after secondary unilateral cleft lip rhinoplasty | Three years
  Use computer software program to compare the nostril symmetry preoperatively and postoperatively: columella height (mm), columella width (mm), nostril height (mm), nostril width (mm), nose base (mm)
Assessment of ratio of the nose in harmony with the face after secondary unilateral cleft lip rhinoplasty | Three years
  Measure the angles and ratios of the nose and its relation to the face (nasal projection and length, Goodle ratio, nasolabial angle)

SECONDARY OUTCOMES:
Objective assessment of functional outcomes | Three years
  Objective measurement will be taken preoperatively and 6 months postoperatively using acoustic rhinometry
Subjective assessment using Rhinoplasty Outcome Evaluation Questionnaire (ROE) | Three years
  Patients will be asked 6 questions from ROE questionnaire preoperatively and postoperatively to assess mental / emotional and quality of life

CONTACTS AND LOCATIONS:
Overall Officials: KieuTho Nguyen, MD, PhD, Study Director — University of Medicine and Pharmacy at Ho Chi Minh City
Locations (1):
- University of Medicine and Pharmacy at HCMC, Ho Chi Minh City, Vietnam